CLINICAL TRIAL: NCT03630237
Title: Distribution of Highly Sensitive Troponin in the Critically Unwell & Associated Mortality. The DIGNITY Study
Brief Title: Distribution of Highly Sensitive Troponin in the Critically Unwell & Associated Mortality
Acronym: DIGNITY
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital Southampton NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: RHM CAR0557
Record Dates: First submitted 2018-08-09; First posted 2018-08-14 (Actual); Last update posted 2019-07-08 (Actual); Status verified 2019-07

CONDITIONS: Myocardial Infarction; Myocardial Injury
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Intensive care population: All patients admitted to any of the three adult intensive care units (general, cardiac & neurosciences) at a large teaching hospital. These patients will have a high sensitivity troponin added onto biochemistry samples requested by the clinical team.

SUMMARY:
The current diagnostic criteria for a heart attack require evaluation of a patient's symptoms and ECG but importantly a blood test called troponin. With advancing technology this test has become more sensitive and is now called a high sensitivity troponin. This is a very effective way of rapidly excluding a heart attack if the test is negative. However there are a number of causes of a raised high sensitivity other than a heart attack, particularly critical illness states. In the absence of features of a heart attack an abnormal result therefore suggests that the heart is inflamed or unwell causing the release of high sensitivity troponin. The DIGNITY study will examine the consequences of high sensitivity troponin elevation in patients in intensive care and assess whether it has a role as a biomarker for predicting outcome.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (aged 18 years or older) admitted to any of the three intensive care facilities on site (general, cardiac and neurosciences)
* Biochemistry samples already taken as part of routine clinical care during the ICU stay

Exclusion Criteria:

* Patients aged less than 18 years
* No biochemistry samples taken within the ICU stay

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive patients admitted any of the three adult intensive care units at a large teaching hospital that have at least one biochemistry sample performed as part of their routine care
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2019-01-28 (Actual); Primary Completion 2019-10-01 (Estimated); Study Completion 2019-10-01 (Estimated)

PRIMARY OUTCOMES:
Association between high sensitivity troponin and inpatient mortality on all patients admitted to each of the ICU environments at a large teaching hospital | During intensive care admission

SECONDARY OUTCOMES:
Distribution of high sensitivity troponin results for different admissions to intensive care | During intensive care admission
  Distribution of high sensitivity troponin results in
  * Medical admissions
  * Trauma / emergency surgical admissions
  * Planned surgical admissions
  * Post cardiac surgical patients
  * Neurosurgical patients
Association between high sensitivity troponin results and duration of ventilation | Within twenty eight days
Association between high sensitivity troponin results and length of intensive care admission | Number of days not in intensive care within twenty eight days of original intensive care admission
Association between high sensitivity troponin results and requirement for inotropic support | During intensive care admission

CONTACTS AND LOCATIONS:
Overall Officials: Nick Curzen, BM, PhD, Principal Investigator — University Hospital Southampton NHS Foundation Trust
Locations (1):
- Univeristy Hospital Southampton, Southampton, United Kingdom

IPD SHARING:
Plan to Share IPD: No